CLINICAL TRIAL: NCT06169644
Title: The Psychological Impact of GTN on Women Who Have Completed Chemotherapy Treatment
Acronym: PI-GTN
Status: Recruiting | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH22800; 331718 (Other: IRAS)
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Gestational Trophoblastic Neoplasia
Keywords: Gestational; Trophoblastic; Disease; Neoplasia; GTD; GTN
MeSH Terms: conditions — Gestational Trophoblastic Disease; Disease; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chemotherapy-treated GTN Patients: Patients with a diagnosis of Gestational Trophoblastic Neoplasia who completed chemotherapy treatment between 6 weeks and 24 months prior to the study. No IMP intervention to be administered, patients to be involved in a qualitative interview.

SUMMARY:
A cross-sectional retrospective study of a sample of 20 women who completed single agent or multi agent chemotherapy: between 6 weeks and 24 months post treatment involving a semi structured telephone interview. A patient sample of 20 is proposed for the study. These are all the patients who meet the inclusion criteria below and are thus eligible for the study. These patients will be contacted via telephone by the principal investigator to inform them of the study and invite participation. A proposed sample size of 20 is sufficient to generate data to address the central questions and furthermore, this sample size is adequate because the intention is to gain insight into the experiences of patients' perceptions about their psychological experiences.

Objectives:

* Gaining insight into the emotional impact of GTN post treatment
* Ascertaining if health professionals are providing adequate psychological support
* Identifying sources of support that patients accessed post completion of treatment
* Identifying potential areas of improvement in the follow up support for future patients

Criteria for inclusion:

* Treated with chemotherapy for a GTN diagnosis
* Completed treatment between 6 weeks and 24 months
* Are able to provide informed consent
* Have no cognitive impairment as judged by the treating clinician

Criteria for exclusion

* Treatment received less than 6 weeks ago
* Treatment received more than 24 months ago
* Non-English speaking

Outcome measures are not appropriate in this qualitative study. However outputs from this study include increasing knowledge and insight into:

* patients' experiences of their psychological experiences post chemotherapy
* patients' perspective of the support received after their treatment
* potential areas of improvements in care

DETAILED DESCRIPTION:
Research question:

What is the psychological impact on women with GTN who have completed chemotherapy treatment?

Objectives:

* Gaining insight into the emotional impact of GTN post treatment
* Ascertaining if health professionals are providing adequate psychological support
* Identifying sources of support that patients accessed post completion of treatment
* Identifying potential areas of improvement in the follow up support for future patients

Abstract:

Gestational Trophoblastic Neoplasia is highly curative but can have psychological consequences for women due to the nature of the diagnosis. Little is known about the psychological impact of diagnosis and treatment experienced by women following the completion of treatment. As the specialist centre for GTN in the North of the UK, it is important to understand the experiences and care needs of our patients. The aim of the study is to explore women's experiences following treatment, how they managed any negative impacts and investigate if there is gap in the follow up support provided to patients after treatment.

The study aims to have 20 participants who received chemotherapy. Semi-structured telephone interviews will be conducted; each interview will be digitally recorded and transcribed verbatim. Thematic analysis will be used to generate in depth descriptions of the patients experiences. The findings will enable health care professionals working closely with this unique group of patients to gain some understanding of the patient perspective; recommendations will be made to improve the support and provision of care these patients receive after their treatment has completed.

Aim:

The aim of the study is to explore the experiences of women with GTN following completion of chemotherapy

Plan of investigation:

Methodology A cross-sectional retrospective study of a sample of 20 women who completed single agent or multi agent chemotherapy: between 6 weeks and 24 months post treatment involving a semi structured telephone interview. This is felt to be appropriate as this topic has received very little research attention for this rare disease and the study aims to capture the patients' own descriptions of their symptoms and experiences. The timeline will capture different perspectives from the varying treatments that patients received, this may provide valuablet insight into patient experiences during different time points.

Telephone interviews will be conducted to gain insight into the patient's experiences. The rationale for using the telephone method is based on the geographical location of our patients. It is not feasible for the investigators to travel to individual homes to conduct the interviews or ask patients to travel. This method has the advantage in that it is relatively inexpensive. The telephone interview offers a robust method of eliciting information from patients about the quality of their care which could help to design improved services. The telephone interviews were designed following discussions with the clinical team and with the aim of answering the research question.

Setting All interviews will be recorded via telephone and take place at Weston Park Hospital. The principal investigator will be responsible for negotiating dates and times of the interview and contacting the participants the day before to ensure they are still available for the scheduled interview. The principal investigator will ensure a designated quiet room is available for the interviews without any interruptions. Each interview will be digitally recorded and transcribed verbatim using an external company- Lawson Hardwick Limited 1st class secretarial services. An hour will be allocated for each interview.

Sample A patient sample of 20 is proposed for the study. These are all the patients who meet the inclusion criteria below and are thus eligible for the study. These patients will be contacted via telephone by the principal investigator to inform them of the study and invite participation. A proposal of 20 is sufficient to generate data to address the central questions and furthermore, this sample size is adequate because the intention is to gain insight into the experiences of patients' perceptions about their psychological experiences.

Criteria for inclusion:

* Treated with chemotherapy for a GTN diagnosis
* Completed treatment between 6 weeks and 24 months
* Are able to provide informed consent
* Have no cognitive impairment as judged by the treating clinician

Criteria for exclusion

* Treatment received less than 6 weeks ago
* Treatment received more than 24 months ago
* Non-English speaking

Recruitment Each of the participants will receive a written information leaflet via email with the details of the nature of study and a written consent form for them to sign and return. The principal investigator will be responsible for contacting the patients once the consent forms have been returned to discuss the study and answer any questions. The interview schedule will be sent prior to the interviews. This will enable them to think about what they would like to say, and importantly, offer them the opportunity to tell their experience in depth.

Intervention:

* Patients are selected as potential participants from the GTN database by the principal investigator
* Patients are contacted by the principal investigation via telephone to invite them to the study
* Patients are emailed the information leaflet along with the written consent form to return back
* If the patients consent to participate in the study the chief investigator will contact participants to discuss
* An interview will be arranged at a time and date convenient to both the patient and the investigator

Outcome measures Outcome measures are not appropriate in this qualitative study. However outputs from this study include increasing knowledge and insight into:

* patients' experiences of their psychological experiences post chemotherapy
* patients' perspective of the support received after their treatment
* potential areas of improvements in care

Analysis Thematic analysis will be used to generate in depth descriptions of the patients experiences. This process of analysis involves looking for themes which are present in the interviews and making comparisons and contrasts between the different respondents. The thematic analysis will be carried out by three investigators. Independent analysis will be carried out separately then meetings will be scheduled to analyse and discuss any agreements and discrepancies to ensure reliability of the interpretations of the data.

Data Collection Data will be collected using telephone semi structured interviews; the interview schedule was developed using the expertise from the research team and on the basis of the aims of the study.

Ethical and safety issues The risks associated with this project are minimal. There are no medical or invasive procedures involved. Therefore, this study does not envisage any harm to be caused to the participant and it is unlikely that the study will encounter any adverse events. It is felt that contacting the patients to invite them to participate is a justified method because the centre has built an excellent rapport with their patients. These patients received treatment at Weston Park Hospital over a number of months; over this period, they have built good trusting relationships with their clinical nurse specialists. Furthermore, these patients continue to be followed up in clinic and via telephone after the treatment has completed. It is possible that the nature of data collection, focusing on personal experiences, may result in some distress to some participants. Both the clinical and research team have extensive experience of caring for patients with cancer. The researchers have relevant experience in working in cancer care and are skilled at talking to patients and will be able to recognise patient distress. If necessary, and with the patients consent, other supportive networks will be made available. The research team will have direct access to the clinical nurse specialist team and be able to refer patients back to their allocated CNS (with the participant's consent).

Patients who agree to participate in the study will be emailed an information sheet explaining the nature of the study and what it entails. Participants will need to sign and return the consent form. It is noted that there may be recall bias as some patients who received treatment almost 24 months ago may not have any symptoms, or not recall in detail compared to those patients who have completed their treatment less than 6 months ago. The use of telephone and email is deemed appropriate as patients often use this method to contact their nursing team and all emails are provided on registration.

There is a potential that during the interview a participant mentions an aspect of care that raises concern regarding care quality, client safety or negligence. If this occurs the study team member will act accordingly, and act follow refer back to the appropriate service provider or care professional.

Subject Withdrawal:

Participants will be able to withdraw from the study at any point; their data will be disposed of using the trust guidelines. If there is sufficient data generated then the study will continue.

Confidentiality All study data including the interview recordings and transcriptions will be identifiable only by an ID number which will be assigned on signing the consent form. Any identifying details will be removed and the transcriptions will be anonymous. The data will be stored securely and confidentially. The interviews will be conducted in a private quiet room. All study data will be stored securely and confidentially in accordance with the Data Protection Act 2018. The data will be kept in locked cupboards and on password protected computers at each of the Trust's centres. The data will be securely kept for future research on the Trust's computer with a secured password.

Involvement of service users:

Two patients who will not be participating in the study have been involved in reviewing the interview questions.

Strategy for taking the work forward if the research project is productive:

The results will be disseminated within the MDT and presented at the next European meeting and International Society for the Study of Trophoblastic Diseases conference in 2024. The findings will enable health care professionals working closely with this unique group of patients to gain some understanding of the patient perspective and importantly improve the patient experience, furthermore, gaining a close insight and improving their own knowledge.

Intellectual property arrangements:

The intellectual property arrangements will be standard for research conducted in the NHS and funded within charitable sources.

End of study definition The study will end when all the data is analysed.

ELIGIBILITY:
Inclusion Criteria:

* Treated with chemotherapy for a GTN diagnosis
* Completed treatment between 6 weeks and 24 months
* Are able to provide informed consent
* Have no cognitive impairment as judged by the treating clinician

Exclusion Criteria:

* Treatment received less than 6 weeks ago
* Treatment received more than 24 months ago
* Non-English speaking

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — GTN affects the female reproductive organs, and as such only those with female biological anatomy. Therefore, only those of female biological sex would meet the eligibility criteria.
Study Population: A patient sample of 20 is proposed for the study. These are all the patients who meet the inclusion criteria and are thus eligible for the study. The patients will have a history of Gestational Trophoblastic Neoplasia, and have received chemotherapy between 6 weeks and 24 months ago, and presented to Weston Park Cancer Centre for this treatment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Common themes of psychological experiences post-chemotherapy | 1 hour interviews
  Thematic analysis will be used to interpret common themes of patient experiences following chemotherapy for GTN
Common opinions of post-treatment support | 1 hour interviews
  Thematic analysis will be used to interpret common patient perspectives of the support received after their treatment
Themes of Suggested Improvement in Patient Care | 1 hour interviews
  Thematic analysis will be used to interpret common suggestions of how patient care can be improved for those receiving chemotherapy for GTN.

CONTACTS AND LOCATIONS:
Overall Officials: Kamaljit Singh, Principal Investigator — Nurse Consultant
Locations (1):
- Weston Park Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No intention to share IPD.

DOCUMENTS (1):
  • Study Protocol (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT06169644/Prot_000.pdf